CLINICAL TRIAL: NCT01717027
Title: Open Label, Single Dose, Randomized, Crossover Study To Evaluate The Pharmacokinetics And Relative Bioavailability Of Oxycodone Following Oral Administration Of 40 Mg Doses Of PF 00345439 Taken Whole Under Fed Conditions And After Chewing Under Fasted Conditions In Healthy Volunteers
Brief Title: Pharmacokinetics And Relative Bioavailability Study Of Oxycodone in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pain Therapeutics (Industry)
Responsible Party: Sponsor
Organization: PainT (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B4501034
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: pharmacokinetics; bioavailability; oxycodone; management of moderate to severe pain
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Experimental): Single dose of 40 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone
- Treatment B (Experimental): Single dose of 40 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone
- Treatment C (Experimental): Single dose of 40 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone
- Treatment D (Experimental): Single dose of 40 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — One capsule of 40 mg PF-00345439 Formulation A, single dose, taken whole and under fed conditions
  Arms: Treatment A
Drug: Oxycodone — One capsule of 40 mg PF-00345439 Formulation J, single dose, taken whole and under fed conditions
  Arms: Treatment B
Drug: Oxycodone — One capsule of 40 mg PF-00345439 Formulation K, single dose, taken whole and under fed conditions
  Arms: Treatment C
Drug: Oxycodone — One capsule of 40 mg PF-00345439 Formulation J or K, single dose, chewed and under fasted conditions
  Arms: Treatment D

SUMMARY:
To estimate the pharmacokinetics and relative bioavailability of oxycodone after administration of 40 mg doses of PF-00345439 formulations taken whole under fed conditions and after chewing under fasted conditions in healthy volunteers

DETAILED DESCRIPTION:
This study will estimate the pharmacokinetics and relative bioavailability of oxycodone following oral administration of single 40 mg doses of PF-00345439 Formulations J and K compared with the reference PF-00345439 Formulation A, all taken whole and under fed conditions in healthy volunteers.

In addition, the study will estimate the pharmacokinetics and relative bioavailability of oxycodone followingoral administration of single 40 mg doses of PF-00345439 Formulation J or K (to beselected based on Periods 1-3) after chewing under fasted conditions compared to that taken whole in the fed state in healthy volunteers, and assess the single-dose safety and tolerability of oxycodone inPF-00345439 formulations in healthy volunteers when administered under a naltrexone block.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between 18 and 55 years of age (inclusive).

Exclusion Criteria:

* Evidence or history of clinically significant disease.
* Positive urine drug test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2012-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) (if data permit, otherwise Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUClast]) of oxycodone. | 0, 0.5, 1, 2, 4, 6, 8, 12, 14, 16, 24, 36, 48 hours post-dose
Maximum Observed Plasma Concentration (Cmax) | 0, 0.5, 1, 2, 4, 6, 8, 12, 14, 16, 24, 36, 48 hours post-dose

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of oxycodone, as data permit | 0, 0.5, 1, 2, 4, 6, 8, 12, 14, 16, 24, 36, 48 hours post-dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) of oxycodone, as data permit. | 0, 0.5, 1, 2, 4, 6, 8, 12, 14, 16, 24, 36, 48 hours post-dose
Plasma Decay Half-Life of oxycodone, as data permit. | 0, 0.5, 1, 2, 4, 6, 8, 12, 14, 16, 24, 36, 48 hours post-dose
Concentration at time 24 hours (C24) of oxycodone, as data permit. | 0, 0.5, 1, 2, 4, 6, 8, 12, 14, 16, 24, 36, 48 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4501034&StudyName=Pharmacokinetics%20And%20Relative%20Bioavailability%20Study%20Of%20Oxycodone%20in%20Healthy%20Volunteers%0A